CLINICAL TRIAL: NCT02836873
Title: A Double Blind Placebo Controlled Study to Evaluate the Effect of Bexagliflozin Tablets on Hemoglobin A1c in Patients With Type 2 Diabetes Mellitus and Moderate Renal Impairment
Brief Title: Safety and Efficacy of Bexagliflozin in Type 2 Diabetes Mellitus Patients With Moderate Renal Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: THR-1442-C-448
Record Dates: First submitted 2016-07-14; First posted 2016-07-19 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — bexagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bexagliflozin tablets, 20 mg (Active Comparator): Each subject will receive a bexagliflozin tablet, 20 mg, once daily for the duration of the study.
  Interventions: Drug: Bexagliflozin
- Placebo tablets (Placebo Comparator): Each subject will receive a placebo (inactive) tablet once daily for the duration of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bexagliflozin — Bexagliflozin tablet, 20 mg
  Other Names: EGT0001442; EGT0001474
  Arms: Bexagliflozin tablets, 20 mg
Drug: Placebo — Placebo (inactive) tablet to match the active comparator
  Arms: Placebo tablets

SUMMARY:
This was a phase 3, multi-center, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of oral administration of bexagliflozin at 20 mg versus placebo in subjects with T2DM, moderate renal impairment and inadequate glycemic control.

DETAILED DESCRIPTION:
The phase 3, double-blind, placebo-controlled parallel-group study was conducted at investigative sites in the US, Japan, France and Spain. Approximately 300 subjects were to be randomly assigned to receive bexagliflozin tablets, 20 mg, or placebo in equal ratio for 24 weeks.

The study was to enrolled male and female participants who had T2DM with an HbA1c between 7.0 and 10.5% (inclusive) and stage 3 chronic kidney disease (CKD) as defined by an eGFR of ≥ 30 and< 60 mL min-1 per 1.73 m2 at the screening visit and one additional time of measurement between 1 and 12 months prior to screening. Subjects were either treatment naïve or were treated with a stable regimen of anti-diabetic medications.

All eligible subjects were to enter a one-week single-blind, placebo run-in period. Subjects who were compliant in taking run-in medication, had screening eGFR ≥ 30 and< 60 mL min-1 per 1.73 m2, and had stable GFR (no more than 20% change in eGFR between a historical value and the value determined at the screening visit) were eligible for randomization. Randomization was stratified by HbA1c level (7.0 to 8.5% or 8.6 to 10.5%), anti-diabetic treatment regimen and eGFR (30 - 44 mL min-1 per 1.73 m2 or 45 - 59 mL min-1 per 1.73 m2). At least 135 subjects in each of the eGFR groups were planned.

Study subjects were to schedule clinic visits at weeks 2, 6, 12, 18, and 24 for safety and efficacy evaluation. At weeks 2 and 18, the visits were to be conducted via phone interviews unless an in-person visit was considered clinically advisable. A final follow-up visit was to be conducted at week 26 or two weeks after the last dose of investigational product if the subject withdrew prior to week 24.

ELIGIBILITY:
Each subject was required to meet the following criteria at the time of enrollment to be eligible for the study:

1. To have been male or non-pregnant female ≥ 20 years of age. Women of childbearing potential were required to agree to use contraception throughout the study to avoid any possible pregnancy. Females who were surgically sterile (hysterectomy, oophorectomy) or postmenopausal (absence of menses for greater than 12 months and age > 45 years) were eligible if they tested negative on the urine pregnancy test.
2. To have had a diagnosis of T2DM with an HbA1c between 7.0 and 10.5% (inclusive) at the time of screening.
3. To have been treatment naïve or to have been treated with a stable regimen of anti-diabetic medications. At the time of screening, the doses and frequency of all anti-diabetic medications were to have been stable for 8 weeks.
4. To have had an eGFR ≥ 30 and < 60 mL min-1 per 1.73 m2 at 2 time points: screening (V1), and 1 additional time point between 1 and 12 months of screening (may be obtained from available medical records). The eGFR was calculated by the MDRD equation.
5. To have had a body mass index (BMI) ≤ 45 kg per m2 (inclusive).
6. To have been taking stable doses of medications for hypertension or hyperlipidemia (if applicable) for at least 30 days prior to randomization
7. To have had stable eGFR between the historic value and day of screening (no more than 20% change in eGFR between the most recent historical value and the value determined at the screening visit V1).

9.3.2 Exclusion Criteria

Potential participants who exhibited any of the following characteristics were excluded from the study:

1. A diagnosis of type 1 diabetes mellitus or maturity-onset diabetes of the young (MODY)
2. A hemoglobinopathy that could affect HbA1c measurement
3. Frequent symptomatic hypoglycemia (greater than one episode per week on average)
4. A history of genitourinary tract infection within 6 weeks of screening or history of ≥ 3 genitourinary infections requiring treatment within the last 6 months
5. A cancer, active or in remission for < 3 years (Non-melanoma skin cancer or basal cell carcinoma or carcinoma in situ of the cervix were not grounds for exclusion)
6. A history of alcohol or illicit drug abuse in the past 2 years
7. Evidence of abnormal liver function tests (total bilirubin or alkaline phosphatase > 1.5 × upper limit of normal (ULN) with the exception of isolated Gilbert's syndrome); or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × ULN
8. A history of MI, stroke or hospitalization for heart failure, or hospitalization for unstable angina in the prior 3 months
9. Evidence of NYHA class IV heart failure at screening or randomization
10. A history of taking an SGLT2 inhibitor within 3 months of screening
11. Any condition, disease, disorder, or clinically relevant laboratory abnormality that, in the opinion of the PI, would jeopardize the subject's appropriate participation in this study or obscure the effects of treatment
12. A current status of pregnancy or breastfeeding
13. A current status of renal replacement therapy (peritoneal or hemodialysis) or a history of renal transplantation
14. A corrected serum calcium < 8 mg dL-1 at screening (V1) or randomization (V3)
15. Uncontrolled hypertension (systolic blood pressure >170 mm Hg or diastolic blood pressure >110 mm Hg)
16. Participation in another interventional trial or exposure to an investigational drug within 30 days or 7 half-lives of screening, whichever was longer
17. Previous exposure to bexagliflozin or EGT0001474
18. Evidence of having skipped dosing more than once during the run-in period
19. A fasting blood glucose value during the run-in period ≥ 250 mg dL-1 (13.9 mmol L-1) associated with severe clinical signs or symptoms of hyperglycemia
20. Any episode of symptomatic hypoglycemia during the run-in period in which symptoms were severe
21. An inability to comprehend or unwillingness to provide written informed consent in accordance with institutional and regulatory guidelines

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Allegretti, M.D., Study Director — Massachusetts General Hospital
Locations (46):
- United States (22):
  - Research Site, Fresno, California
  - Research Site, La Palma, California
  - Research Site, Lincoln, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Dimas, California
  - Research Site, Monument, Colorado
  - Research Site, Norwalk, Connecticut
  - Research Site, Hollywood, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Paducah, Kentucky
  - Research Site, Auburn, Maine
  - Research Site, Rockport, Maine
  - Research Site, Nashua, New Hampshire
  - Research Site, The Bronx, New York
  - Research Site, Stow, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Austin, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, Round Rock, Texas
  - Research Site, San Antonio, Texas
- France (5):
  - Research Site, Dijon
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Vénissieux
- Japan (13):
  - Research Site, Atsugi-shi, Kanagawa
  - Research Site, Kamakura-shi, Kanagawa
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Kawagoe-shi, Saitama
  - Research Site, Kawaguchi-shi, Saitama
  - Research site, Sayama-shi, Saitama
  - Research Site, Hachioji-shi, Tokyo
  - Research Site, Minato-ku, Tokyo
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Toshima-ku, Toyko
- Spain (6):
  - Research Site, Alcalá de Henares
  - Research Site, Alicante
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818

RESULTS

PARTICIPANT FLOW:
Groups:
- Bexagliflozin 20 mg: Each subject will receive a bexagliflozin tablet, 20 mg, once daily for the duration of the study.
- Placebo: Each subject will receive a placebo (inactive) tablet once daily for the duration of the study.
Period: Overall Study
Arm/Group | Bexagliflozin 20 mg | Placebo
Started | 157 | 155
Completed | 152 | 144
Not Completed | 5 | 11
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bexagliflozin 20 mg | Placebo | Total
Number analyzed (Participants) | 157 | 155 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (8.36) | 69.9 (8.29) | 69.6 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 51 | 116
  Male | 92 | 104 | 196
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 17 | 24
  Not Hispanic or Latino | 149 | 138 | 287
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 61 | 59 | 120
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 9 | 6 | 15
  White | 83 | 88 | 171
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 53 | 50 | 103
  Japan | 58 | 58 | 116
  France | 12 | 16 | 28
  Spain | 34 | 31 | 65
Height [Mean (Standard Deviation); unit: cm] | 164.8 (9.94) | 164.7 (10.58) | 164.8 (10.25)
Body Weight [Mean (Standard Deviation); unit: kg] | 82.90 (20.509) | 82.59 (21.196) | 82.75 (20.820)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.29 (5.988) | 30.10 (5.774) | 30.20 (5.874)
SBP Categories [Count of Participants; unit: Participants]
  < 130 mm Hg | 50 | 42 | 92
  > 130 mm Hg | 107 | 113 | 220
eGFR in Sub-group [Mean (Standard Deviation); unit: mL/min/1.73 m^2]
  Stage 3a CKD: eGFR High Group | 51.76 (5.307) | 51.27 (4.404) | 51.52 (4.884)
  Stage 3b CKD: eGFR Low Group | 37.79 (4.572) | 37.87 (4.629) | 37.83 (4.586)
Subjects in eGFR Sub-group at Baseline [Count of Participants; unit: Participants]
  Stage 3a CKD: eGFR High Group | 86 | 80 | 166
  Stage 3b CKD: eGFR Low Group | 71 | 75 | 146

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at 24 Weeks
Description: The primary efficacy objective of this trial is to evaluate the placebo-adjusted change in HbA1c from baseline after 24 weeks of treatment with 20 mg bexagliflozin tablets in type 2 diabetic subjects with moderate renal impairment.
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Bexagliflozin 20 mg | Placebo
Number analyzed (Participants) | 157 | 155
percentage of glycated hemoglobin | -0.59 (0.065) | -0.31 (0.066)
Statistical Analysis 1: Comparison: Bexagliflozin 20 mg vs Placebo; This is a mixed-effects repeated measures analysis including region, screening anti-diabetic treatment regimen, baseline eGFR, treatment, visit, treatment-by-visit interaction and baseline HbA1c as a fixed effect covariate. Data from Weeks 6, 12, and 24 are used in the model; Test type: Superiority; p = 0.0026, Mixed-effects repeated measures; Region, screening anti-diabetic treatment, baseline eGFR, treatment, visit, treatment-by-visit and baseline HbA1c value as fixed effect covariates; Difference of LS Means = -0.28, 95% CI 2-sided [-0.46 to -0.10]

2. Secondary Outcome: Change in Body Weight From Baseline to Week 24 in Subjects With a BMI ≥ 25 kg/m2
Description: A secondary objective is to evaluate the effect of bexagliflozin 20 mg on the placebo-adjusted change in BMI from baseline to week 24 in subjects with a BMI ≥ 25 kg/m2.
Time Frame: 24 weeks
Population: Only number of subjects with a value at baseline and at the specific visit is included.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Bexagliflozin 20 mg | Placebo
Number analyzed (Participants) | 122 | 117
kg | -2.31 (0.265) | -0.55 (0.269)
Statistical Analysis 1: Comparison: Bexagliflozin 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed-effects repeated measures; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -1.76, 95% CI 2-sided [-2.50 to -1.03]

3. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) in Subjects With Baseline SBP ≥ 130 mm Hg at Week 24
Description: A secondary objective is to evaluate the effect of bexagliflozin 20 mg on the placebo-adjusted change from baseline in SBP to in subjects with baseline SBP ≥ 130 mm Hg at Week 24.
Time Frame: 24 weeks
Population: Only number of subjects with a value at baseline and at Week 24 is included.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bexagliflozin 20 mg | Placebo
Number analyzed (Participants) | 104 | 108
mm Hg | -10.14 (1.477) | -7.51 (1.460)
Statistical Analysis 1: Comparison: Bexagliflozin 20 mg vs Placebo; Test type: Superiority; p = 0.2035, Mixed-effects repeated measures; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -2.63, 95% CI 2-sided [-6.70 to 1.44]

4. Secondary Outcome: Change From Baseline in HbA1c in Subjects With Stage 3a CKD (eGFR 45 to 59 mL/Min/1.73 m2) at Week 24
Description: A secondary objective is to evaluate the effect of bexagliflozin 20 mg on the placebo-adjusted change in HbA1c from baseline in subjects with stage 3a CKD (eGFR 45 to 59 mL/min/1.73 m2) at week 24.
Time Frame: 24 weeks
Population: Subjects who had the eGFR between 45 and 59 mL/min/1.73 m2 are included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Bexagliflozin 20 mg | Placebo
Number analyzed (Participants) | 86 | 80
percentage of glycated hemoglobin | -0.63 (0.086) | -0.44 (0.089)
Statistical Analysis 1: Comparison: Bexagliflozin 20 mg vs Placebo; Test type: Superiority; p = 0.1156, Mixed-effects repeated measures; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.20, 95% CI 2-sided [-0.44 to 0.05]

5. Secondary Outcome: Change From Baseline in HbA1c in Subjects With Stage 3b CKD (eGFR 30 to 44 mL/Min/1.73 m2) at Week 24
Description: A secondary objective is to evaluate the effect of bexagliflozin 20 mg on the placebo-adjusted change in HbA1c from baseline in subjects with stage 3b CKD (eGFR 30 to 44 mL/min/1.73 m2) at week 24.
Time Frame: 24 weeks
Population: Subjects with eGFR between 30 and 44 mL/min/1.73 m2 were included in this anlaysis.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycated hemoglobin
Arm/Group | Bexagliflozin 20 mg | Placebo
Number analyzed (Participants) | 71 | 75
percentage of glycated hemoglobin | -0.57 (0.100) | -0.20 (0.097)
Statistical Analysis 1: Comparison: Bexagliflozin 20 mg vs Placebo; Test type: Superiority; p = 0.0078, Mixed-effects repeated measures; [statistical method as in outcome 1, analysis 1]; Difference of LS Means = -0.37, 95% CI 2-sided [-0.65 to -0.10]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Week -1 (Visit 2) to Week 26 (Visit 29).
Arm/Group | Bexagliflozin 20 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/155
Serious Adverse Events (participants affected / at risk) | 11/157 | 9/155
Other Adverse Events (participants affected / at risk) | 56/157 | 42/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bexagliflozin 20 mg (N=157) | Placebo (N=155)
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Intestinal ischemia (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Adenocarcinoma colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathic anthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexagliflozin 20 mg (N=157) | Placebo (N=155)
Polyuria (Renal and urinary disorders) | 12 (15) | 7 (7)
Acute kidney injury (Renal and urinary disorders) | 8 (9) | 6 (6)
Nasopharyngitis (Infections and infestations) | 11 (13) | 13 (21)
Urinary tract infection (Infections and infestations) | 10 (12) | 5 (5)
Bronchitis (Infections and infestations) | 8 (8) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 5 (5)
Nausea (Gastrointestinal disorders) | 8 (9) | 11 (12)
Hypoglycaemia (Metabolism and nutrition disorders) | 40 (258) | 40 (261)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI has no right to publish the trial results.

DOCUMENTS (2):
  • Study Protocol (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT02836873/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT02836873/SAP_001.pdf